CLINICAL TRIAL: NCT02111512
Title: Phase 4 Study to Assess the Safety of Nasal Influenza Immunisation in Egg Allergic Children - a Multicentre Observational Study
Brief Title: Safety of Nasal Influenza Immunisation in Egg Allergic Children - The SNIFFLE 2 Study
Acronym: SNIFFLE-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); Public Health England (Other Government)
Responsible Party: Principal Investigator, Paul Turner, MRC Clinician Scientist, Imperial College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHM CHI 0714; 2014-001537-92 (EudraCT Number); 17189 (Registry Identifier: UKCRN)
Record Dates: First submitted 2014-04-04; First posted 2014-04-11 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Egg Hypersensitivity
MeSH Terms: conditions — Egg Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Egg allergic children (Other): Children with a physician diagnosis of egg allergy will be recruited to receive the intranasal LAIV as part of a safety surveillance study
  Interventions: Drug: Administration of Live attenuated influenza vaccine (LAIV)

INTERVENTIONS:
Drug: Administration of Live attenuated influenza vaccine (LAIV)

SUMMARY:
Egg allergy is common in early childhood, affecting at least one in 50 preschool children. Influenza ("'flu") vaccines contain egg protein, as the vaccine is cultured in hen's eggs. There is robust data to support the safety of influenza vaccines (containing low or negligible amounts of egg protein) in patients with egg allergy.

A new influenza vaccine, known as LAIV (Live Attenuated Intranasal Vaccine) has recently been approved by a number of licensing boards and is given by a spray into the nose. This new vaccine has been available in the United States for several years and is highly effective and against influenza infection, with an excellent safety profile in children without egg allergy. However, LAIV is also grown in hen's eggs and contains egg protein, and there are NO published data on the safety of LAIV in egg-allergic children. In SNIFFLE 1 Study, 433 doses were given to 282 egg-allergic children; data is currently being analysed.

The objective of this multicentre study is to further assess the safety of intranasal LAIV in egg-allergic children, in order to demonstrate that these children can safely be given the new LAIV within a primary care health environment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 - 17 years old
* Physician-diagnosis of egg allergy

Exclusion Criteria:

1. Clinical resolution of egg allergy
2. Contraindications to LAIV (notwithstanding allergy to egg protein):

   * Hypersensitivity to the active ingredients, gelatin or gentamicin (a possible trace residue)
   * Previous systemic allergic reaction to LAIV
   * Previous allergic reaction to an influenza vaccine (not LAIV) is a relative contra-indication, which must be discussed with the site PI to confirm patient suitability
   * Children/adolescents who are clinically immunodeficient due to conditions or immunosuppressive therapy such as: acute and chronic leukaemias; lymphoma; symptomatic HIV infection; cellular immune deficiencies; and high-dose corticosteroids. NB: LAIV is not contraindicated for use in individuals with asymptomatic HIV infection; or individuals who are receiving topical/inhaled corticosteroids or low-dose systemic corticosteroids or those receiving corticosteroids as replacement therapy, e.g. for adrenal insufficiency.
   * Children and adolescents younger than 18 years of age receiving salicylate therapy because of the association of Reye's syndrome with salicylates and wild-type influenza infection.
3. Contraindication to vaccination on that occasion, due to child being acutely unwell:

   * Febrile ≥38.0oC in last 72 hours
   * Acute wheeze in last 72 hours requiring treatment beyond that normally prescribed for regular use by the child's treating healthcare professional
   * Recent admission to hospital in last 2 weeks for acute asthma
   * Current oral steroid for asthma exacerbation or course completed within last 2 weeks

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 779 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of allergic reaction to nasal influenza vaccination using a Live Attenuated Influenza Vaccine (LAIV) in egg-allergic children | Within 2 hours of vaccine administration

SECONDARY OUTCOMES:
Incidence of delayed symptoms up to 72 hours after nasal influenza vaccination with LAIV in egg-allergic children | 72 hours after vaccine administration
Asthma control test | 4 weeks post LAIV
  To assess for a change in asthma control (by validated questionnaire) pre and 4 weeks post LAIV immunisation.

OTHER OUTCOMES:
Incidence of immediate allergic reaction to LAIV in the subgroups described below. | Within 2 hours of vaccine administration
  1. By age group 2-5, 6-11, 12-17 years
  2. Children with a clinician-assessed history of reaction to egg in the previous 12 months
  3. Children with evidence of >95% likelihood of egg allergy (as per published criteria) within the past 3 months
  4. Children with evidence of >95% likelihood of egg allergy (as per published criteria) within the past 12 months
  5. children with a previous history of anaphylaxis to egg protein
  6. children who have reacted previously to airborne traces of egg
  7. children who have egg allergy but are tolerant of baked egg
  8. Children who have previously received influenza vaccine
  9. Presence of physician-diagnosed asthma / recurrent wheeze

CONTACTS AND LOCATIONS:
Overall Officials: Mich Erlewyn-Lajeunesse, DM FRCPCH, Principal Investigator — University Hospitals Southampton NHS Foundation Trust; Paul J Turner, FRACP PhD, Principal Investigator — Imperial College London
Locations (29):
- United Kingdom (29):
  - Ulster Hospital, Belfast, Northern Ireland
  - Royal United Hospital Bath NHS Trust, Bath
  - Sandwell General Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Hospital for Sick Children, Edinburgh
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth
  - Wye Valley NHS Trust, Hereford
  - Cambridgeshire Community Services NHS Trust (Hinchingbrooke Hospital), Huntingdon
  - Leeds Children's Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's Hospital, Liverpool
  - Barts Health NHS Trust, London
  - Evelina Children's Hospital, London
  - Imperial College Healthcare NHS Trust (St. Mary's Hospital), London
  - Kings College Hospital NHS Foundation Trust, London
  - London St George's Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Luton and Dunstable Hospital, Luton
  - Manchester Royal Children's, Manchester
  - Newcastle Freeman Hospital, Newcastle
  - Oxford, Oxford
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Sheffield Children's Hospital NHS Foundation Trust, Sheffield
  - Shrewsbury and Telford Hospital NHS Trust, Shrewsbury
  - University Hospitals Southampton NHS Foundation Trust, Southampton
  - Warrington & Halton Hospitals NHS Foundation Trust, Warrington
  - Hampshire Hospital NHS Foundation Trust, Winchester

REFERENCES:
- [Result] Turner PJ, Southern J, Andrews NJ, Miller E, Erlewyn-Lajeunesse M; SNIFFLE-2 Study Investigators. Safety of live attenuated influenza vaccine in young people with egg allergy: multicentre prospective cohort study. BMJ. 2015 Dec 8;351:h6291. doi: 10.1136/bmj.h6291. PMID 26645895